CLINICAL TRIAL: NCT02132234
Title: Effects of Biological Treatment on Blood Pressure and Endothelial Function in Patients With Rheumatoid Arthritis, Psoriatic Arthritis and Ankylosing Spondylitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Collaborators: Departmet of Rheumatology, J Dietl Hospital, Krakow, Poland (Unknown)
Responsible Party: Principal Investigator, Tomasz Guzik, MD, PhD, Jagiellonian University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UJ-KChWiMWsi-Reu
Record Dates: First submitted 2014-04-28; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-05

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis; Ankylosing Spondylitis; Hypertension
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Spondylitis, Ankylosing; Hypertension | interventions — Etanercept; Adalimumab; Certolizumab Pegol; Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Biological treatment (Experimental): Patients with high disease activity receiving biological treatment according to rheumatologic indication:
  * etanercept 50 mg s.c. every week
  * adalimumab 40 mg s.c. every 2 weeks
  * certolizumab 400 mg s.c. every 2 weeks for 4 weeks, then 200mg every 2 weeks
  * infliximab 3 or 5 mg/kg i.v. 2 and 6 weeks from the first admission, then every 8 weeks
  Interventions: Drug: Etanercept; Drug: Adalimumab; Drug: Certolizumab; Drug: Infliximab
- control group (Placebo Comparator): Patients with high disease activity receiving other than biological treatment and receiving placebo.

INTERVENTIONS:
Drug: Etanercept — biological treatment according to rheumatologic indication
  Arms: Biological treatment
Drug: Adalimumab — biological treatment according to rheumatologic indication
  Arms: Biological treatment
Drug: Certolizumab — biological treatment according to rheumatologic indication
  Arms: Biological treatment
Drug: Infliximab — biological treatment according to rheumatologic indication
  Arms: Biological treatment

SUMMARY:
The aim of this study is to evaluate the influence of anti tumor necrosis factor-alpha (TNF-α) treatment on blood pressure, endothelial function and immune cell phenotype in patients with rheumatoid arthritis, psoriatic arthritis and ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

For patients suffering from rheumatoid arthritis:

* rheumatoid arthritis diagnosed based on The American Rheumatism Association Criteria from 1987
* ineffective treatment with 2 disease-modifying antirheumatic drugs (DMARDs) for 6 months each, including treatment with maximal doses of methotrexate for at least 3 months (or intolerance to treatment)
* high disease activity - Disease Activity Score 28 (DAS 28) > 5,1 measured twice, with a 1-month interval
* for patients with mainly lower limbs affected with DAS 28 > 3,7

For patients suffering from Ankylosing Spondylitis:

* Ankylosing Spondylitis diagnosed based on Modified New York Criteria
* ineffective treatment with 2 non-steroidal anti-inflammatory drugs (administered separately) in maximal recommended or maximal tolerated dose for 3 months
* high disease activity -Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) > 4 measured twice, with a 12-week interval
* spinal pain > 4cm on 10cm Visual Analogue Scale (VAS) measured twice, with a 12-week interval
* general disease activity assessment > 5 (0-10 scale) performed after the 2nd VAS and BASDAI assessment

For patients suffering from Psoriatic Arthritis:

- Psoriatic arthritis diagnosed based on the Bennett or Classification Criteria for Psoriatic Arthritis (CASPAR Criteria)

If peripheral joints are affected:

active disease assessed twice, with a 4-week interval on stable treatment, after 2 DMARDs treatment for at least 4 months

Criteria of active disease (all have to be met):

* At least 5 out of 66 joints swollen - assessed twice, with a 4-week interval
* At least 5 out of 68 joints tender - assessed twice, with a 4-week interval
* general disease activity assessment of 4 or 5 in the Likert scale (0- 5 scale) performed by patient
* general disease activity assessment of 4 or 5 in the Likert scale (0- 5 scale) performed by physician
* general disease activity assessment > 5 (0-10 scale) performed after 2nd assessment of number of tender and swollen joints

If axial joints are affected:

* Sacroiliac joints affected according to the New York Criteria of Ankylosing Spondylitis
* Active and severe disease assessed twice, with a 12-week interval, stable treatment, ineffective treatment with 2 nonsteroidal anti-inflammatory drugs (administered separately) in maximal recommended or maximal tolerated dose for 3 months each

Criteria of active disease (all must be present):

* BASDAI > 4 measured twice, with a 12-week interval
* spinal pain > 4cm on 10 cm in the VAS measured twice, with a 12-week interval
* general disease activity assessment > 5 (0-10 scale) Patients can take steroid in stable dose within one month - maximal dose 10mg/day of prednisone.

Exclusion Criteria:

* non-consenting patient
* pregnancy
* breast-feeding
* allergy for the drug or any component
* cardiac insufficiency (NYHA III or IV)
* active infection
* infection within the last 3 months: hepatitis, pneumonia, pyelonephritis
* opportunistic infection within the last 2 months: active infection of cytomegalovirus, Pneumocystis carinii
* joint infection within the last 12 months
* endoprosthesis infection within the last 12 months or any time if the joint was not replaced
* exacerbation of lung-, kidney-, liver- or heart insufficiency during treatment
* demyelinating disease or its symptoms
* pancytopenia or aplastic anemia
* pre-cancer stage
* neoplasm within the last 5 years including solid tumors and neoplasm of haematopoietic or lymphatic system with risk of recurrence or progression
* active alcoholic disease
* chronic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in blood pressure | prior to receiving anti-TNF-α treatment, 12 weeks
  Ambulatory Blood Pressure Monitoring (ABPM)

SECONDARY OUTCOMES:
Change from baseline in endothelial function | prior to receiving anti-TNF-α treatment, 12 weeks
  Flow Mediated Dilatation / Endo Pat

OTHER OUTCOMES:
Changes in immune cell subset populations from baseline | prior to receiving anti-TNF-α treatment, 12 weeks
  determination of subsets, activation markers, intracellular cytokine production

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Guzik, MD, PhD, Study Chair — Jagiellonian University; Bogdan Batko, MD, PhD, Study Chair — Department of Rheumatology, J. Dietl Hospital, Krakow, Poland
Locations (1):
- Katedra Chorób Wewnętrznych i Medycyny Wsi, Uniwersytet Jagielloński, Krakow, Skarbowa 4, Poland